CLINICAL TRIAL: NCT00198939
Title: Neurological Influences on Drug Prevention Intervention
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 5R01DA015075-03 (NIH); 5R01DA015075-03 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Youths At-risk for Drug Use/Abuse
Keywords: drug prevention; adolescence; middle school; randomized trial; family therapy; cognitive-behavioral; efficacy; selected youth; indicated youth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Psychoeducation (Active Comparator): Drug education curriculum was delivered to participants assigned to this condition.
  Interventions: Other: Psychoeducation
- Conitive Behavorial Therapy (Experimental): The cognitive-behavioral program introduces youths to problem-solving behavior change principles and study skills to promote school achievement.
  Interventions: Behavioral: Integrated Family and Cognitive-Behavioral Drug Prevention Intervention
- Family Therapy (Experimental): Participants assigned to the Family Therapy arm received a family-centered intervention to support targeted adolescent behavior change. The family therapy component of IFCBT includes engagement, active treatment, and maintenance phases.
  Interventions: Behavioral: Integrated Family and Cognitive-Behavioral Drug Prevention Intervention
- Intergrated Family and Cognitve Behavioral Therapy (Experimental): Participants assigned to the IFCBT arm received the Cognitive Behavioral Therapy and Family Therapy intervention components.
  Interventions: Behavioral: Integrated Family and Cognitive-Behavioral Drug Prevention Intervention

INTERVENTIONS:
Behavioral: Integrated Family and Cognitive-Behavioral Drug Prevention Intervention — The family therapy component of IFCBT includes engagement, active treatment, and maintenance phases. The cognitive program focuses on harmful effects of drugs and strategies to better manage drug abuse risks. The cognitive-behavioral program introduces youths to problem-solving behavior change principles and study skills to promote school achievement.
  Arms: Conitive Behavorial Therapy; Family Therapy; Intergrated Family and Cognitve Behavioral Therapy
Other: Psychoeducation — Drug education curriculum was delivered to participants assigned to this condition.
  Arms: Psychoeducation

SUMMARY:
In this R01 study, a randomized clinical trial is proposed to evaluate the efficacy of a drug abuse prevention intervention for indicated middle school youth that coordinates family and teen-based components. The Family Management Intervention is comprised of a parent-focused curriculum to foster parenting skills followed by brief family therapy to foster adaptive family communication and age-appropriate roles. The Teen Achievement Intervention is comprised of a clinician-delivered learning strategy curriculum to foster academic achievement followed by a similar yet peer-facilitated curriculum to foster self-efficacy and prosocial peer networks. In the first study aim, we seek to evaluate the separate and possibly synergistic effects of the Family Management and Teen Achievement components on post intervention drug use, problem behavior, psychological distress, and academic achievement of indicated youth. Innovative analytic strategies are subsequently used to elucidate mediated pathways by which the interventions might reduce drug involvement and problem behavior by promoting changes in targeted skills and behavior change processes. The possibility of effect-modification also is considered, with a focus on neurocognitive, internalizing/externalizing, and demographic factors, in an effort to discern why interventions work for some youth but not others. This application revision has sought to address well-taken concerns cited by the reviewers while maintaining proposal strengths. In response to a key limitation, this revision includes further specification of anticipated relationships between neurocognitive variables, skill acquisition levels, and prevention intervention outcomes among indicated youth. Study hypotheses on specific neurocognitive effects are informed by empirical findings and the clinical experience of investigative team members specializing in neuropsychology. If successful, this project should improve prevention practices by identifying malleable behavior change processes fostered by effective interventions. Improving our understanding of how individual characteristics of indicated youth, such as neurocognitive deficits or externalizing problems, influence the development of skills during interventions and subsequent outcomes may also help to improve existing prevention interventions. The significance of the proposed study is underscored further by the substantial size of the targeted population of indicated youth, and the range of morbidities and mortality that often result when early warning signs of drug abuse are not addressed.

ELIGIBILITY:
Inclusion Criteria:

* 11 to 15 year old middle school students

Exclusion Criteria:

* Acute suicidal, homicidal, psychotic ideation
* Problem severity indicating outpatient or residential treatment

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2005-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Alcohol use abstinence and frequency | 3, 6, 9, 12, and 18 month Follow-up assement
  Personal Experience Inventory (PEI) is a youth self-report drug use inventory that assesses the frequency and quantity of substance use and drug abuse risk factors, such as deviant behavior and peer drug use.
Marijuana use abstinence and frequency | 3, 6, 9, 12, and 18 Month Follow-up Assessment
  The Personal Experience Inventory (PEI) is a youth self-report drug use inventory that assesses the frequency and quantity of substance use and drug abuse risk factors, such as deviant behavior and peer drug use.
Other drug use abstinence and frequency | 3, 6, 9, 12, 18 month Follow-up Assessment
  The Adolescent Stage of Change Scale (ASCS) consists of items to measure youths' motivation to change drug use behavior. Urine will also be analyzed for the presence of drugs, such as cannabinoids, cocaine, opiates, amphetamine, methamphetamine, MDMA, benzodiazepines, and barbiturates using gas chromatography/mass spectrometry methods.

SECONDARY OUTCOMES:
Academic achievement | 3,6,9,12, and 18 month assessment
  The Interview on Sociodemographic Characteristics is administered to collect information on grades, academic achievement, days truant, school behavior problems, detention, suspension, and expulsion.
Family functioning | 3,6,9,12, and 18 month follow-up assessment
  The Family Assessment Measure (FAM) is a self-report tool for parents and children that measures change processes targeted by the family systems component of IFCBT, including appropriate role performance, parental control, and communication.
Learning Strategy Skill | 3,6,9,12, and 18 month assessment
  The Motivated Strategies for Learning Questionnaire (MSLQ) assesses adolescents' motivation to learn in school and use of effective learning strategies that are addressed during the Learning Strategy Training module of IFCBT.
Legal Involvement | 3,6,9, 12, and 18 month follow-up assessment
  The parent and adolescent versions of the Missouri Assessment for Genetics Interview for Children (MAGIC) address diagnostic symptoms associated with DSM-IV criteria including conduct disorder and antisocial personality disorder and includes questions on legal involvement.

CONTACTS AND LOCATIONS:
Overall Officials: William W. Latimer, PhD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Latimer WW, Winters KC, D'Zurilla T, Nichols M. Integrated family and cognitive-behavioral therapy for adolescent substance abusers: a stage I efficacy study. Drug Alcohol Depend. 2003 Sep 10;71(3):303-17. doi: 10.1016/s0376-8716(03)00171-6. PMID 12957348